CLINICAL TRIAL: NCT05538806
Title: TTFields in General Routine Clinical Care in Patients With Pleural Mesothelioma Study - TIGER Meso Study
Brief Title: TTFields in General Routine Clinical Care in Patients With Pleural Mesothelioma Study
Acronym: TIGER Meso
Status: Recruiting | Type: Observational
Sponsor: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP-RS-001
Record Dates: First submitted 2022-09-06; First posted 2022-09-14 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2024-12

CONDITIONS: Pleural Mesothelioma
Keywords: Pleural Mesothelioma; TTFields
MeSH Terms: conditions — Mesothelioma, Malignant

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group 1: all patients will receive routine clinical care and TTFields
  Interventions: Device: TTFields

INTERVENTIONS:
Device: TTFields — all patients will receive routine clinical care and TTFields

SUMMARY:
The purpose of this post-authorisation medical device study is to obtain real life data on the use of Tumor Treating Fields (TTFields) in patients with pleural mesothelioma in routine clinical care. Patients with pleural mesothelioma and clinical indication for TTFields treatment will be enrolled in the study after signing Informed consent to use their data and process it centrally for research purposes. The clinical indication for TTFields is one of the inclusion criteria and is defined prior to inclusion by the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Histologically confirmed pleural mesothelioma without any option of curative resection
* Planned treatment with NovoTTF-200T System according to IFU and medical guidelines
* Life expectancy more than 3 months at day of enrollment
* Signed informed consent for use and processing of data

Exclusion Criteria:

• Previous treatment with NovoTTF-200T for more than 1 week at day of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, histologically confirmed pleural mesothelioma without any option of curative resection
Sampling Method: Non-Probability Sample
Enrollment: 198 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Time from diagnosis of pleural mesothelioma to death of any cause as median overall survival time. | 54 Months

SECONDARY OUTCOMES:
Number of TTFields treatment-related SAEs, as assessed by the CEC, within total observation period, standardized to average annual incidences. | 3 years + 18 months follow up
Changes in quality of life comparing baseline with 3 and 6 months after start of TTFields therapy. | QoL will be assessed at baseline, 3 and 6 months.

CONTACTS AND LOCATIONS:
Locations (23):
- Germany (20):
  - Lungenklinik Gauting, Gauting, Bavaria
  - University Hospital Regensburg, Regensburg, Bavaria
  - Klinikum Bremen-Ost, Bremen, City state Bremen
  - Asklepios Klinikum Harburg, Harburg, Hamburg
  - University Medicine Göttingen, Göttingen, Lower Saxony
  - University Hospital Carl Gustav Carus Dresden, Dresden, Saxony
  - Charité Universitätsmedizin Berlin, Berlin
  - Lungenklinik Heckeshorn, Berlin
  - Kliniken der Stadt Koeln, Cologne
  - Florence-Nightingale-Hospital, Düsseldorf
  - Klinikum Essen-Mitte, Essen
  - University Hospital Essen, Essen
  - Niels-Stensen Hospital, Georgsmarienhütte
  - Krankenhaus Martha-Maria Halle-Doelau, Halle
  - Medizinische Hochschule Hannover, Hanover
  - Lungenklinik Hemer, Hemer
  - Evangelisches Krankenhaus Herne, Herne
  - Krankenhaus Bethanien Moers, Moers
  - GEHO Muenster, Münster
  - Fachkliniken Wangen, Wangen
- Italy (2):
  - Azienda Ospedaliero-Universitaria di Alessandria "SS. Antonio e Biagio e C. Arrigo", Alessandria
  - Humanitas Gavazzeni, Bergamo
- Erasmus MC Cancer Centre, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided